CLINICAL TRIAL: NCT02641379
Title: Randomized, Multicenter Study to Find Optimal Treatment Duration in Patients With Chronic Hepatitis C and Subtype 1 or 4 Depending on HCV RNA Level at Week 8 and Week 12
Brief Title: A Study of Peginterferon Alfa-2a (Pegasys) When Administered in Combination With Ribavirin in Patients With Chronic Hepatitis C (CHC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17131
Record Dates: First submitted 2015-12-11; First posted 2015-12-29 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (4):
- PEG-IFN 24 weeks (Experimental): Participants will receive PEG-IFN (180 microgram [mcg]), subcutaneously (sc), once weekly for 24 weeks and Ribavirin 1000-1200 milligram per day (mg/day) (<75 kilogram (kg); >75 kg) for 24 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- PEG-IFN 24/72 weeks (Experimental): Participants will receive PEG-IFN (180 mcg), sc, once weekly and Ribavirin 1000-1200 mg/day (<75kg; >75 kg) till week 24; if patient is still HCV RNA positive. Treatment will be stopped if participant is HCV RNA negative at week 24 -treatment with PEG-IFN (180 mcg), sc, once weekly and Ribavirin 1000-1200 mg/day (<75kg; >75 kg) till week 72
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- PEG-IFN 48 weeks (Experimental): Participants will receive PEG-IFN (180 mcg), sc, once weekly for 48 weeks and Ribavirin 1000-1200 mg/day (<75kg; >75 kg) for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- PEG-IFN 72 weeks (Experimental): Participants will receive PEG-IFN (180 mcg), sc, once weekly for 72 weeks and Ribavirin 1000-1200 mg/day (<75 kg; > 75 kg) for 72 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — PEG-IFN is available as 180 microgram (mcg) per 0.5 mL, prefilled syringe and pen for single dose sc. injection\n
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin is available as 200 mg tablets

SUMMARY:
This study will compare the efficacy and safety of 2 different treatment durations of peginterferon alfa-2a (Pegasys) plus ribavirin in patients with CHC. The anticipated time on study treatment is 1-2 years, and the target sample size is greater than (>) 500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with chronic hepatitis C and genotype 1 (1a or 1b) or genotype 4
* Age between 18 and 70 years
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Present with at least one elevated serum alanine-aminotransferase (ALT) level higher than normal in the last 6 months before therapy start including the screening period
* Positive HCV-RNA level in serum
* Laboratory parameters (within 35 days prior to study start): -Hepatitis A anti - IgM negativity, HIV-Ab negativity, HBsAg negativity, Hemoglobin values > 12 g/dl in women or > 13 g/dl in men, Leukocyte count (WBC) > 3 000 /mcl, Platelets count > 100 000/mcl, Creatinine not 1.5 times higher than normal, normal TSH, normal uric acid with a maximum tolerance of 15 % in patients without history of gout
* Liver biopsy findings within 6 months prior to study therapy consistent with the diagnosis of chronic hepatitis C infection with or without compensated cirrhosis. Biopsies older than 1 year are eligible only after direct communication with the principal investigator
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug. If there is no laboratory report existing, the physician should make an entry in the medical history that the pregnancy test was negative.
* All fertile females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end. All fertile men with female partners must be using two forms of effective contraception during treatment and during the 7 months after treatment end.
* Written informed consent obtained

Exclusion Criteria:

* Any IFN and / or Pegylated IFN and ribavirin therapy at any previous time
* Class B or C cirrhosis as coded by Child Pugh classification
* Women with ongoing pregnancy or breast feeding
* Therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug
* Any investigational drug 6 weeks prior to the first dose of study drug
* Drug addiction within 1 year prior to study start (patients participating in an official methadone program are eligible)
* Diabetes mellitus in patients receiving an insulin therapy
* Hemophiliac patients (due to the increased risk of requested liver biopsy)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease. Exception: if there is a current psychiatric report which certifies there is no contraindication to interferon therapy, patient may be included
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis etc.)
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of a severe seizure disorder or current anticonvulsant use
* History of severe cardiac disease and severe coronary heart disease within the last 6 months (angina pectoris, congestive heart failure, recent myocardial infarction, severe hypertension or significant arrhythmia). If there is clinical suspicion of coronary heart disease cardiologic workup of the patient prior to study entry is recommended.
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* History or other evidence of severe illness, malignancy or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of major organ transplantation with an existing functional graft
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Inability or unwillingness to provide informed consent or abide by the requirements of the study

Additional exclusion criteria concerning ribavirin:

* Male partners of women who are pregnant
* Any patient with an increased baseline risk for anemia (e.g. thalassemia, spherocytosis, history of GI bleeding, etc) or for whom anemia would be medically problematic
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL would not be well-tolerated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2003-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (14):
- Austria (14):
  - Feldkirch
  - Gratwein
  - Graz
  - Innsbruck
  - Krems
  - Linz
  - Oberndorf
  - Oberpullendorf
  - Ried-innkreis
  - Salzburg
  - Vienna
  - Villach
  - Wels
  - Wiener Neustadt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 2 parts. Part 1 was conducted from 16 May 2003 to 12 September 2008 at 21 centers in Austria; Part 2 of this study was conducted from 19 October 2009 to 15 November 2013 at 15 centers in Austria.
Pre-assignment Details: A total of 545 participants were enrolled in Part 1, of which 5 participants were treated but were not included in any analysis population due to a missing post-baseline safety assessment. A total of 176 participants were enrolled in Part 2 of this study.
Groups:
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1): Eligible participants received pegylated interferon alpha-2a (PEG-IFN alfa-2a) at a dose of 180 microgram (mcg) subcutaneously (SC) once weekly for a total of 48 weeks and ribavirin at a dose of 1,000 milligram/day (mg/day) [for participants with a body weight </= 75 kilogram (kg)] or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants were randomized to Group A based on the presence of an early virological response (EVR) defined as non-detectable serum hepatitis C virus ribonucleic acid (HCV RNA) [< 600 international units/milliliter (IU/ml)] by quantitative polymerase chain reaction (PCR) or a 2-log10 decrease or greater compared to baseline serum HCV RNA, shortly after Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for 48 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 72 weeks. After Week 48, participants were administered a lower dose of PEG-IFN alfa-2a of 135 mcg/week until Week 72. Participants were randomized to Group B based on the presence of an EVR defined as non-detectable serum HCV RNA (< 600 IU/ml) by quantitative PCR or a 2-log10 decrease or greater compared to baseline in serum HCV RNA by quantitative PCR, shortly after Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally; initially for 24 weeks. Participants without an EVR at Week 12 (< 2-log10 decrease in HCV RNA as compared with baseline) were assigned to Group C and received treatment until Week 24. If HCV RNA became non-detectable at Week 24 then treatment was continued for a total of 72 weeks. Participants were administered a lower dose of PEG-IFN alfa-2a after Week 48 (135 mcg/week, until Week 72). Participants with detectable HCV RNA (≥ 50 IU/ml) at Week 24 were required to discontinue treatment. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 24 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 24 weeks. Participants with a rapid virological response (RVR) at Week 4 of treatment [HCV RNA level, <50 IU/ml by qualitative PCR assay, COBAS Amplicor HCV Test, version 2.0] were assigned to Group D. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin (Not Randomized) (Part 1): Eligible participants who were not randomized to any treatment group in Part 1 of the study were included in this group. These participants were a part of the safety analysis population which included participants who received at least on dose of (either) the study drug (PEG-IFN alfa-2a and/or ribavirin) and had at least one post-baseline safety assessment.
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants were randomized to Group A1 if they showed positive HCV RNA level (≥ 15 IU/ml, TaqMan® HCV Test) at Week 4 and at Week 8, a negative HCV RNA level or > 2-log10 decline (TaqMan HCV test) at Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 72 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 72 weeks. Participants were randomized to Group B1 if they showed positive HCV RNA level (≥ 15 IU/ml, TaqMan® HCV Test) at Week 4 and at Week 8, a negative HCV RNA level or > 2-log10 decline (TaqMan HCV test) at Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally; initially for 24 weeks. Participants without a > 2-log10 drop of HCV RNA level at Week 12 were assigned to Group C (Part 2). For participants who were HCV RNA-positive at Week 24, treatment was stopped. For participants who were negative for HCV RNA at Week 24, treatment was continued for a total of 72 weeks. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 24 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 24 weeks. Participants with a negative HCV-RNA level at Week 4 (< 15 IU/ml, TaqMan HCV Test) were assigned to Group D. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and also received ribavirin at a dosage of 1,000 mg/day (for participants with a body weight ≤ 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants with a positive HCV RNA level at Week 4 (≥ 15 IU/ml, TaqMan HCV Test) and negative HCV RNA level at Week 8 (≤ 15 IU/ml, TaqMan HCV Test) were assigned to Group E. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin (Not Assigned) (Part 2): Eligible participants who were not assigned to any treatment group in Part 2 were included in this group. These participants were a part of the safety analysis population which included all participants who received at least on dose of (either) study drug (PEG-IFN alfa-2a and/or ribavirin) and had at least one post-baseline safety assessment.
Period: Overall Study
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1) | PEG-IFN Alfa-2a + Ribavirin (Not Randomized) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2) | PEG-IFN Alfa-2a + Ribavirin (Not Assigned) (Part 2)
Started | 142 | 152 | 78 | 156 | 17 | 36 | 25 | 20 | 42 | 45 | 8
Completed | 107 | 101 | 7 | 139 | 0 | 20 | 12 | 1 | 36 | 36 | 0
Not Completed | 35 | 51 | 71 | 17 | 17 | 16 | 13 | 19 | 6 | 9 | 8
Not completed — Exclusion criterion during screening | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of informed consent | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 8 | 2 | 2 | 5 | 1 | 5 | 0 | 1 | 1 | 5
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 5 | 0 | 0 | 0
Not completed — Participant unable to attend study visit | 4 | 10 | 1 | 2 | 5 | 1 | 1 | 1 | 0 | 2 | 0
Not completed — Participant's compliance | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1
Not completed — Participant cannot be reached | 4 | 4 | 0 | 8 | 2 | 1 | 0 | 1 | 0 | 2 | 1
Not completed — PCR positive at Week 24 | 15 | 21 | 62 | 0 | 0 | 6 | 3 | 8 | 0 | 1 | 0
Not completed — PCR positive at follow up 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant showed relapse | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant stopped study/treatment | 1 | 3 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Therapy stopped due to misunderstanding | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Financial problems | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PCR positive at Week 68 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PCR positive at Week 48 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PCR not performed at Week 12 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No PCR at baseline | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PCR positive at Week 28 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PCR sample for Week 4 not drawn | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion criteria not fulfilled | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Baseline viral load unavailable | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Blood could not be drawn | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participation in sili rescue study | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Source data not found | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant showed weight reduction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Non-response Week 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — No 2 Log drop at Week 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Negative PCR result | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant's PCR high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant treated after Week 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Missing PCR result at Week 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — PCR positive | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the safety population which included all participants who received at least on dose of (either) study drug and had at least one post-baseline safety assessment.
Groups:
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants were randomized to Group A based on the presence of an EVR defined as non-detectable serum HCV RNA (< 600 IU/ml) by quantitative PCR or a 2-log10 decrease or greater compared to baseline serum HCV RNA, shortly after Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally; initially for 24 weeks. Participants without an EVR at Week 12 (< 2-log10 decrease in HCV RNA as compared with baseline) were assigned to Group C and received treatment until Week 24. If HCV RNA became non-detectable at Week 24 then treatment was continued for a total of 72 weeks. Participants were administered a lower dose of PEG-IFN alfa-2a after Week 48 (135 mcg/week, until Week 72). Participants with detectable HCV RNA (>= 50 IU/ml) at Week 24 were required to discontinue treatment. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 24 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 24 weeks. Participants with a RVR at Week 4 of treatment [HCV RNA level, <50 IU/ml by qualitative PCR assay, COBAS Amplicor HCV Test, version 2.0] were assigned to Group D. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants were randomized to Group A1 if they showed positive HCV RNA level (>/= 15 IU/ml, TaqMan HCV Test) at Week 4 and at Week 8, a negative HCV RNA level or > 2-log10 decline (TaqMan HCV test) at Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 72 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 72 weeks. Participants were randomized to Group B1 if they showed positive HCV RNA level (>/= 15 IU/ml, TaqMan HCV Test) at Week 4 and at Week 8, a negative HCV RNA level or > 2-log10 decline (TaqMan HCV test) at Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2): Eligible participants received PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and also received ribavirin at a dosage of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants with a positive HCV RNA level at Week 4 (>/= 15 IU/ml, TaqMan HCV Test) and negative HCV RNA level at Week 8 (</= 15 IU/ml, TaqMan HCV Test) were assigned to Group E. Participants had a treatment-free follow-up period of 24 weeks.
- Total: Total of all reporting groups
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1) | PEG-IFN Alfa-2a + Ribavirin (Not Randomized) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2) | PEG-IFN Alfa-2a + Ribavirin (Not Assigned) (Part 2) | Total
Number analyzed (Participants) | 142 | 152 | 78 | 156 | 12 | 36 | 25 | 20 | 42 | 45 | 8 | 716
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (10.7) | 44.2 (10.2) | 46.6 (9.0) | 40.5 (11.7) | 46.5 (9.5) | 44.6 (9.1) | 47.3 (9.8) | 46.6 (8.7) | 37.8 (11.1) | 41.1 (10.2) | 43.6 (15.4) | 43.5 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 53 | 21 | 57 | 4 | 8 | 8 | 5 | 17 | 20 | 3 | 246
  Male | 92 | 99 | 57 | 99 | 8 | 28 | 17 | 15 | 25 | 25 | 5 | 470

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapse Rate in Groups A and B by Genotype at the End of Follow-up (Part 1)
Description: Relapse rate (RR) was defined as the percentage of participants with non-detectable HCV RNA (< 100 copies/ml) at the end of treatment and detectable HCV RNA at the end of follow-up. End of treatment was defined as Week 48 for Group A and Week 72 for Group B, respectively. The end of follow-up was defined as Week 72 for Group A and Week 96 for Group B, respectively. Relapse rate for treatment Groups A and B, stratified for genotype (Genotype I and Genotype IV) and Week 4 response (< 600 units/milliliter [U/ml] and >= 600 U/ml) is presented.
Time Frame: Up to Week 96
Population: The ITT population included all participants randomized and allocated to receive treatments. Here, 'n' = number of participants analyzed according to genotype and Week 4 response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for 48 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 72 weeks. After Week 48, participants were administered a lower dose of PEG-IFN alfa-2a of 135 mcg/week until Week 72. Participants were randomized to Group B based on the presence of an EVR defined as non-detectable serum HCV RNA (< 600 IU/ml) by quantitative PCR or a 2-log10 decrease or greater compared to baseline in serum HCV RNA by quantitative PCR, shortly after Week 12. Participants had a treatment-free follow-up period of 24 weeks.
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1)
Number analyzed (Participants) | 142 | 152
Percentage of participants
  Genotype I, Week 4 response < 600 U/ml,n= 130, 136 | 22.0 [10.6 to 37.6] | 8.3 [1.8 to 22.5]
  Genotype I,Week 4 response >=600 U/ml, n =130, 136 | 52.7 [38.8 to 66.3] | 30.0 [17.9 to 44.6]
  Genotype IV, Week 4 response < 600 U/ml, n =12, 16 | 0.0 [0.0 to 52.2] | 42.9 [9.9 to 81.6]
  Genotype IV, Week 4 response >=600 U/ml, n =12, 16 | 80.0 [28.4 to 99.5] | 80.0 [28.4 to 99.5]
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) vs PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1); For Genotype I, Week 4 response < 600 U/ml: Comparison of Group A versus Group B was carried out using the Chi-Square test; Test type: Superiority or Other; p = 0.1002, Chi-squared
Statistical Analysis 2: Comparison: PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) vs PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1); For Genotype I, Week 4 response >= 600 U/ml: Comparison of Group A versus Group B was carried out using the Chi-Square test; Test type: Superiority or Other; p = 0.0184, Chi-squared
Statistical Analysis 3: Comparison: PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) vs PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1); For Genotype IV, Week 4 response < 600 U/ml: Comparison of Group A versus Group B was carried out using the Chi-Square test; Test type: Superiority or Other; p = 0.0910, Chi-squared
Statistical Analysis 4: Comparison: PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) vs PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1); For Genotype IV, Week 4 response >= 600 U/ml: Comparison of Group A versus Group B was carried out using the Chi-Square test; Test type: Superiority or Other; p = 1.0000, Chi-squared

2. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response in Groups A1, B1, and E by Genotype at the End of Follow-up (Part 2)
Description: The Sustained Virological Response (SVR) was defined as the percentage of participants in each group with non-detectable HCV RNA result at 24 weeks post completion of the treatment period (HCV RNA < 15 IU/ml at Week 72 of Groups A1 and E, and at Week 96 of Group B1). Participants without a HCV RNA results at this time point were considered as non-responders. The end of follow-up was defined as Week 72 for Groups A1 and E, and Week 96 for Group B1. The SVR for treatment Groups A1 + B1 and E, stratified for genotype (Genotype I and Genotype IV) is presented.
Time Frame: Up to Week 96
Population: The ITT population included all participants randomized and allocated to receive treatments. Here, 'n' = the number of participants analyzed according to genotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PEG-IFN Alfa 2a + Ribavirin 48 Weeks (Group A1) (Part 2): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants were randomized to Group A1 if they showed positive HCV RNA level (>/= 15 IU/ml, TaqMan HCV Test) at Week 4 and at Week 8, a negative HCV RNA level or > 2-log10 decline (TaqMan HCV test) at Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa 2a + Ribavirin 72 Weeks (Group B1) (Part 2): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 72 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 72 weeks. Participants were randomized to Group B1 if they showed positive HCV RNA level (>/= 15 IU/ml, TaqMan HCV Test) at Week 4 and at Week 8, a negative HCV RNA level or > 2-log10 decline (TaqMan HCV test) at Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and also received ribavirin at a dosage of 1,000 mg/day (for participants with a body weight ≤ 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants with a positive HCV RNA level at Week 4 (≥ 15 IU/ml) and negative HCV RNA level at Week 8 (≤ 15 IU/ml) were assigned to group E. Participants had a treatment-free follow-up period of 24 weeks.
Arm/Group | PEG-IFN Alfa 2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa 2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2)
Number analyzed (Participants) | 33 | 23 | 45
Percentage of participants
  Genotype I, n = 33, 23, 39 | 30.3 [15.6 to 48.7] | 34.8 [16.4 to 57.3] | 64.1 [47.2 to 78.8]
  Genotype IV, n = 3, 2, 6 | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 84.2] | 50.0 [11.8 to 88.2]
Statistical Analysis 1: Comparison: PEG-IFN Alfa 2a + Ribavirin 48 Weeks (Group A1) (Part 2) vs PEG-IFN Alfa 2a + Ribavirin 72 Weeks (Group B1) (Part 2) vs PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2); Comparison of Groups A1+B1 versus group E stratified by genotype I; Test type: Superiority or Other; p = 0.0021, Cochran-Mantel-Haenszel — The SVR rate i.e., 32.1% participants with genotype I who achieved SVR with 95 % confidence interval of 20.3 to 46.0 in groups A1+B1 was compared with SVR rate in group E using Cochran-Mantel-Haenszel method
Statistical Analysis 2: Comparison: PEG-IFN Alfa 2a + Ribavirin 48 Weeks (Group A1) (Part 2) vs PEG-IFN Alfa 2a + Ribavirin 72 Weeks (Group B1) (Part 2) vs PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2); Comparison of Groups A1+B1 versus group E stratified by genotype IV; Test type: Superiority or Other; p = 0.3031, Cochran-Mantel-Haenszel — The SVR rate i.e., 20.0% participants with genotype IV who achieved SVR with 95 % confidence interval of 0.5 to 71.6 in groups A1+B1 was compared with SVR rate in group E using Cochran-Mantel-Haenszel method

3. Secondary Outcome: Percentage of Participants With Virological Response Rate in Groups A, B, C, and D at the End of Treatment Period (Part 1)
Description: End of treatment response (ETR) rate was defined as the percentage of participants in each group with non-detectable HCV RNA at completion of the treatment period (HCV negative at Week 24 of Group D, Week 48 of Group A and at Week 72 of Groups B and C). Participants without a HCV RNA results at this time point were considered as non-responders. End of the treatment period was defined as Week 48 for Group A, Week 72 for Groups B and C, and Week 24 for Group D.
Time Frame: Up to Week 72
Population: The ITT population included all participants randomized and allocated to receive treatments.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally; initially for 24 weeks. Participants without an EVR at Week 12 (< 2-log10 decrease in HCV RNA as compared with baseline) were assigned to Group C and received treatment until Week 24. If HCV RNA became non-detectable at Week 24 then treatment was continued for a total of 72 weeks. Participants were administered a lower dose of PEG-IFN alfa-2a after Week 48 (135 mcg/week, until Week 72). Participants with detectable HCV RNA (>= 50 IU/ml) at Week 24 were required to discontinue treatment. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 24 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 24 weeks. Participants with a RVR at Week 4 of treatment [HCV RNA level, <50 IU/ml by qualitative PCR assay, COBAS Amplicor HCV Test, version 2.0] were assigned to Group D. Participants had a treatment-free follow-up period of 24 weeks.
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1)
Number analyzed (Participants) | 142 | 152 | 78 | 156
Percentage of participants | 74.6 [66.7 to 81.6] | 64.5 [56.3 to 72.1] | 9.0 [3.7 to 17.6] | 92.3 [86.9 to 96.0]

4. Secondary Outcome: Percentage of Participants Achieving Sustained Virological Response in Groups A, B, C, and D at the End of Follow-up (Part 1)
Description: The SVR was defined as the percentage of participants in each group with a non-detectable HCV RNA result at 24 weeks post-completion of the treatment period (HCV RNA < 15 IU/ml at Week 48 of Group D, at Week 72 of Group A, and at Week 96 of Groups B and C). Participants without a HCV RNA PCR at this time point were considered as non-responders in this calculation. The end of follow-up was defined as Week 72 for Group A, Week 96 for Groups B and C, and Week 48 for Group D.
Time Frame: Up to Week 96
Population: The ITT population included all participants randomized and allocated to receive treatments.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1)
Number analyzed (Participants) | 142 | 152 | 78 | 156
Percentage of participants | 45.1 [36.7 to 53.6] | 48.0 [39.9 to 56.3] | 6.4 [2.1 to 14.3] | 73.7 [66.1 to 80.4]

5. Secondary Outcome: Mean Short Form-36 Questionnaire Scores for Groups A and B Over Time (Part 1)
Description: The Short Form-36 (SF-36) is a quality of life instrument consisting of a 36-item questionnaire. The SF-36 items were scored and transformed according to the SF-36 Health Survey Manual and Interpretation Guide. Summary scores for SF-36 dimensions (physical functioning, role functioning, bodily pain, general health, vitality, social functioning, mental health, health transition) as well as physical and mental summary measures were compiled after imputation of mean scores for missing items if more than 50% of dimension-related items were available. Scores for health transition ranged from 0 (worst) to 5 (best). Scores for all other dimensions ranged from 0 (worst) to 100 (best). The mean SF-36 scores are presented at Baseline (Day 1), Week 24, Week 48, Week 72 (for Groups A and B) and at Week 96 (for Group B). Lower score indicate worsening.
Time Frame: Baseline (Day 1), Week 24, Week 48, Week 72, and Week 96
Population: The ITT population included all participants randomized and allocated to receive treatments. Here, 'n' = the number of participants analyzed at a given time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1)
Number analyzed (Participants) | 106 | 123
scores on a scale
  Physical Functioning, Baseline, n = 106, 121 | 86.9 (15.1) | 87.0 (17.8)
  Physical Functioning, Week 24, n = 77, 90 | 61.8 (28.2) | 69.2 (22.6)
  Physical Functioning, Week 48, n = 67, 77 | 66.1 (26.2) | 66.8 (23.1)
  Physical Functioning, Week 72, n = 65, 68 | 89.8 (14.1) | 70.3 (24.6)
  Physical Functioning, Week 96, n = 0, 59 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 87.0 (20.4)
  Role Functioning - Physical, Baseline,n = 105, 120 | 74.7 (36.3) | 76.2 (36.9)
  Role Functioning - Physical, Week 24, n = 77, 88 | 39.0 (43.0) | 45.7 (41.9)
  Role Functioning - Physical, Week 48, n = 66, 76 | 40.7 (39.9) | 42.2 (44.0)
  Role Functioning - Physical, Week 72, n = 65, 67 | 81.5 (32.9) | 47.4 (43.5)
  Role Functioning - Physical, Week 96, n = 0, 58 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 84.5 (29.9)
  Bodily Pain, Baseline, n = 103, 120 | 82.3 (22.5) | 83.5 (22.9)
  Bodily Pain, Week 24, n = 76, 91 | 68.2 (31.1) | 70.0 (29.6)
  Bodily Pain, Week 48, n = 67, 77 | 69.5 (28.6) | 66.8 (30.6)
  Bodily Pain, Week 72, n = 64, 70 | 85.4 (23.2) | 67.3 (29.3)
  Bodily Pain, Week 96, n = 0, 61 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 90.2 (19.8)
  General Health, Baseline, n = 102, 119 | 64.5 (17.9) | 66.3 (19.7)
  General Health, Week 24, n = 75, 83 | 58.9 (19.0) | 55.1 (22.8)
  General Health, Week 48, n = 63, 74 | 58.1 (20.2) | 56.3 (19.2)
  General Health, Week 72, n = 65, 62 | 71.7 (18.8) | 60.1 (19.3)
  General Health, Week 96, n = 0, 59 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 70.3 (18.5)
  Vitality, Baseline, n = 103, 116 | 56.8 (20.9) | 58.9 (22.5)
  Vitality, Week 24, n = 75, 88 | 40.3 (24.0) | 40.6 (23.6)
  Vitality, Week 48, n = 66, 77 | 40.6 (23.8) | 41.2 (21.2)
  Vitality, Week 72, n = 63, 67 | 66.9 (18.9) | 43.5 (22.4)
  Vitality, Week 96, n = 0, 59 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 62.9 (21.1)
  Social Functioning, Baseline, n = 105, 121 | 79.8 (21.9) | 81.6 (22.0)
  Social Functioning, Week 24, n = 77, 91 | 64.4 (28.5) | 64.1 (30.3)
  Social Functioning, Week 48, n = 67, 78 | 71.6 (24.0) | 57.2 (27.5)
  Social Functioning, Week 72, n = 65, 70 | 86.3 (22.3) | 63.8 (29.4)
  Social Functioning, Week 96, n = 0, 61 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 83.4 (23.4)
  Role Functioning - Emotional,Baseline,n = 104, 120 | 71.5 (39.3) | 75.8 (36.6)
  Role Functioning - Emotional, Week 24, n = 76, 88 | 36.8 (42.4) | 43.9 (43.3)
  Role Functioning - Emotional, Week 48, n = 66, 74 | 41.7 (41.0) | 42.8 (42.9)
  Role Functioning - Emotional, Week 72, n = 65, 66 | 80.5 (32.8) | 43.4 (43.4)
  Role Functioning - Emotional, Week 96, n = 0, 58 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 84.5 (31.4)
  Mental Health, Baseline, n = 103, 115 | 69.6 (18.7) | 71.9 (19.1)
  Mental Health, Week 24, n = 76, 88 | 60.7 (19.3) | 57.9 (21.5)
  Mental Health, Week 48, n = 66, 77 | 62.6 (19.8) | 59.6 (20.7)
  Mental Health, Week 72, n = 63, 67 | 76.3 (16.2) | 60.8 (18.5)
  Mental Health, Week 96, n = 0, 59 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 72.3 (14.6)
  Reported Health Transition, Baseline, n = 105, 123 | 3.1 (0.9) | 3.0 (0.9)
  Reported Health Transition, Week 24, n = 77, 90 | 3.5 (1.2) | 3.2 (1.2)
  Reported Health Transition, Week 48, n = 67, 77 | 3.2 (1.3) | 3.0 (1.3)
  Reported Health Transition, Week 72, n = 65, 69 | 1.6 (0.9) | 2.3 (1.1)
  Reported Health Transition, Week 96, n = 0, 61 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 1.3 (0.7)

6. Secondary Outcome: Mean Fatigue Severity Scale Scores for Groups A and B Over Time (Part 1)
Description: The Fatigue Severity Scale (FSS) is an instrument consisting of 10 self-administered questions. The FSS items were scored by calculating the average response to all answered items (including the 9 questions and the fatigue symptoms). Each of the 9 questions had answers within a score range of 1-7. A score of 1 for any question indicates less fatigue in everyday life and a score of 7 indicates a higher likelihood of fatigue in everyday life. The mean FSS scores are presented at Baseline (Day 1), Week 24, Week 48 and Week 72 (for Groups A and B) and at Week 96 (for Group B).
Time Frame: Baseline (Day 1), Week 24, Week 48 and Week 72, and Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1)
Number analyzed (Participants) | 104 | 114
scores on a scale
  Baseline, n = 104, 114 | 3.6 (1.5) | 3.4 (1.7)
  Week 24, n = 69, 77 | 4.5 (1.7) | 4.7 (1.7)
  Week 48, n = 59, 63 | 4.7 (1.6) | 4.7 (1.5)
  Week 72, n = 58, 62 | 3.0 (1.5) | 4.3 (1.8)
  Week 96, n = 0, 57 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 3.4 (1.5)

7. Secondary Outcome: Number of Participants With Fibrosis Grades 0 to 4 at Baseline (Part 1)
Description: Liver fibrosis stage was scored using the METAVIR system (Grade 0 to 4). Grade 0 indicates no fibrosis, Grade 1 indicates stellate enlargement of portal tract but without septa formation, Grade 2 indicates enlargement of portal tract with rare septa formation, Grade 3 indicates numerous septa without cirrhosis and grade 4 indicates cirrhosis. The number of participants with fibrosis grades ranging from 0 to 4 at Baseline is presented.
Time Frame: Baseline (Day 1)
Population: The safety population included all participants who received at least on dose of (either) study drug and had at least one post-baseline safety assessment.
Measure: Number; unit: Number of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1) | PEG-IFN Alfa-2a + Ribavirin (Not Randomized) (Part 1)
Number analyzed (Participants) | 142 | 152 | 77 | 156 | 11
Number of participants
  Grade 0 | 11 | 15 | 8 | 17 | 1
  Grade 1 | 38 | 40 | 20 | 57 | 1
  Grade 2 | 64 | 68 | 23 | 58 | 6
  Grade 3 | 18 | 13 | 15 | 10 | 3
  Grade 4 | 11 | 16 | 11 | 14 | 0

8. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events (Part 1)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 96
Population: as for outcome 7
Measure: Number; unit: Number of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1) | PEG-IFN Alfa-2a + Ribavirin (Not Randomized) (Part 1)
Number analyzed (Participants) | 142 | 152 | 78 | 156 | 12
Number of participants
  Number of participants with any AE | 140 | 149 | 76 | 153 | 10
  Number of participants with any SAE | 22 | 28 | 8 | 14 | 2

9. Secondary Outcome: Percentage of Participants With Relapse Rates in Groups A1 and B1 at the End of Follow-up (Part 2)
Description: Virological relapse rate was defined as percentage of participants with non-detectable HCV RNA (< 15 IU/ml) at the EoT and detectable HCV RNA (≥ 15 IU/ml) at the end of FU. The end of treatment was defined as Week 48 in Group A1 and Week 72 in Group B1 and the end of follow-up was defined as Week 72 in Group A1 and Week 96 in Group B1.
Time Frame: Up to Week 96
Population: The ITT population included all participants randomized and allocated to receive treatments.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants were randomized to Group A1 if they showed positive HCV RNA level (>/= 15 IU/ml, TaqMan HCV Test) at Week 4 and at Week 8, a negative HCV RNA level or > 2-log10 decline (TaqMan HCV test) at Week 12. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 72 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 72 weeks. Participants were randomized to Group B1 if they showed positive HCV RNA level (>/= 15 IU/ml, TaqMan HCV Test) at Week 4 and at Week 8, a negative HCV RNA level or > 2-log10 decline (TaqMan HCV test) at Week 12. Participants had a treatment-free follow-up period of 24 weeks.
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2)
Number analyzed (Participants) | 36 | 25
Percentage of participants | 41.2 [18.4 to 67.1] | 38.5 [13.9 to 68.4]

10. Secondary Outcome: Percentage of Participants With Virological Response Rates in Group A1, B1, C and D at the End of the Treatment Period (Part 2)
Description: ETR virological response rate at the end of treatment period was defined as the percentage of participants in each group with non-detectable HCV RNA at completion of the treatment period (HCV RNA quantitative PCR result < 15 IU/ml at Week 24 for Group D, at Week 48 for Group A1, at Week 72 for Groups B1 and C). Participants without a HCV RNA PCR (missing values) at this time point were considered as non-responders in this calculation. The end of treatment period was defined as Week 48 for Group A1, Week 72 for Groups B1 and C1, and Week 24 for Group D.
Time Frame: Up to Week 72
Population: The ITT population included all participants randomized and allocated to receive treatments.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally; initially for 24 weeks. Participants without a > 2-log10 drop of HCV RNA level at Week 12 were assigned to Group C (Part 2). For participants who were HCV RNA-positive at Week 24, treatment was stopped. For participants who were negative for HCV RNA at Week 24, treatment was continued for a total of 72 weeks. Participants had a treatment-free follow-up period of 24 weeks.
- PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 24 weeks and also received ribavirin at a dose of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 24 weeks. Participants with a negative HCV-RNA level at Week 4 (< 15 IU/ml, TaqMan HCV Test) were assigned to Group D. Participants had a treatment-free follow-up period of 24 weeks.
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2)
Number analyzed (Participants) | 36 | 25 | 20 | 42
Percentage of participants | 47.2 [30.4 to 64.5] | 52.0 [31.3 to 72.2] | 5.0 [0.1 to 24.9] | 90.5 [77.4 to 97.3]

11. Secondary Outcome: Percentage of Participants Achieving Sustained Virological Response in Groups C and D by Genotype at the End of Follow-up (Part 2)
Description: The SVR was defined as the percentage of participants in each group with non-detectable HCV RNA result at 24 weeks post completion of the treatment period (HCV RNA < 15 IU/ml at Week 48 of Group D and at Week 96 of Group C). Participants without a HCV RNA results at this time point were considered as non-responders. The end of follow-up was defined as Week 96 for Group C and Week 48 for Group D.
Time Frame: Up to Week 96
Population: The ITT population included all participants randomized and allocated to receive treatments.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2)
Number analyzed (Participants) | 20 | 42
Percentage of participants | 0.0 [0.0 to 16.8] | 73.8 [58.0 to 86.1]

12. Secondary Outcome: Mean Short Form-36 Questionnaire Scores for Groups A1, B1, and C Over Time (Part 2)
Description: The SF-36 is a quality of life instrument consisting of a 36-item questionnaire. The SF-36 items were scored and transformed according to the SF-36 Health Survey Manual & Interpretation Guide. Summary scores for SF-36 dimensions (physical functioning, role functioning, bodily pain, general health, vitality, social functioning, mental health, health transition) as well as physical and mental summary measures were compiled after imputation of mean scores for missing items if more than 50% of dimension-related items were available. Scores for health transition ranged from 0 (worst) to 5 (best). Scores for all other dimensions ranged from 0 (worst) to 100 (best). The mean SF-36 scores were presented at Baseline (Day 1), Week 24, Week 48, Week 72 (for Groups A1, B1 and C) and at Week 96 (for Groups B1 and C). Lower score indicate worsening.
Time Frame: Baseline (Day 1), Week 24, Week 48, Week 72, and Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2)
Number analyzed (Participants) | 22 | 19 | 15
scores on a scale
  Physical functioning, Baseline, n = 22, 18, 15 | 82.5 (22.5) | 83.1 (17.7) | 78.5 (28.8)
  Physical functioning, Week 24, n = 17, 13, 9 | 61.8 (25.8) | 51.2 (25.2) | 72.2 (24.9)
  Physical functioning, Week 48, n = 13, 8, 0 | 66.5 (22.8) | 76.3 (19.8) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Physical functioning, Week 72, n = 10, 7, 1 | 77.0 (18.4) | 80.7 (9.3) | 45.0 (NA) — Data is available only for one participant. Therefore, there is no standard deviation.
  Physical functioning, Week 96, n = 0, 6, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 85.8 (17.7) | NA (NA) — No participants were available for analysis in this arm at Week 96.
  Role Functioning- Physical, Baseline,n =22, 18, 15 | 75.0 (33.6) | 62.0 (42.1) | 53.3 (41.0)
  Role Functioning - Physical, Week 24, n= 17, 13, 8 | 41.2 (44.1) | 15.4 (33.1) | 43.8 (43.8)
  Role Functioning - Physical, Week 48, n = 13, 8, 0 | 41.0 (41.3) | 56.3 (39.5) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Role Functioning - Physical,, Week 72, n= 10, 7,1 | 60.0 (47.4) | 82.1 (37.4) | 0.0 (0.0)
  Role Functioning - Physical, Week 96, n = 0, 5, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 70.0 (32.6) | NA (NA) — No participants were available for analysis in this arm at Week 96.
  Bodily Pain, Baseline, n = 21, 19, 15 | 75.3 (26.7) | 76.3 (25.5) | 66.5 (31.7)
  Bodily Pain, Week 24, n = 17, 13, 8 | 57.9 (28.5) | 45.9 (27.9) | 54.9 (17.8)
  Bodily Pain, Week 48, n = 13, 8, 0 | 66.4 (31.6) | 54.6 (19.2) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Bodily Pain, Week 72, n = 10, 7, 1 | 71.1 (30.1) | 70.4 (15.0) | 62.0 (NA) — Data is available only for one participant. Therefore, there is no standard deviation.
  Bodily Pain, Week 96, n = 0, 6, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 74.5 (19.3) | NA (NA) — No participants were available for analysis in this arm at Week 96.
  General Health, Baseline, n = 22, 16, 14 | 61.8 (18.8) | 56.7 (21.7) | 53.4 (19.1)
  General Health, Week 24, n = 17, 11, 8 | 52.8 (23.6) | 37.1 (14.1) | 57.1 (24.4)
  General Health, Week 48, n = 12, 8, 0 | 54.4 (21.0) | 56.3 (23.8) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  General Health, Week 72, n = 10, 7, 1 | 55.0 (21.8) | 59.9 (16.5) | 35.0 (NA) — Data is available only for one participant. Therefore, there is no standard deviation.
  General Health, Week 96, n = 0, 6, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 52.8 (18.8) | NA (NA) — No participants were available for analysis in this arm at Week 96.
  Vitality, Baseline, n = 21, 18, 15 | 54.0 (21.9) | 52.5 (19.3) | 45.0 (16.0)
  Vitality, Week 24, n = 17, 11, 8 | 37.8 (13.9) | 31.2 (21.7) | 43.1 (17.9)
  Vitality, Week 48, n = 13, 8, 0 | 43.2 (22.1) | 48.1 (17.3) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Vitality, Week 72, n = 9, 7, 1 | 47.2 (23.1) | 60.2 (16.7) | 40.0 (NA) — Data is available only for one participant. Therefore, there is no standard deviation.
  Vitality, Week 96, n = 0, 6, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 56.9 (15.1) | NA (NA) — No participants were available for analysis in this arm at Week 96.
  Social Functioning, Baseline, n = 22, 19, 15 | 84.7 (18.5) | 78.9 (25.0) | 72.5 (33.5)
  Social Functioning, Week 24, n = 17, 13, 8 | 64.7 (26.6) | 56.7 (23.2) | 65.6 (23.9)
  Social Functioning, Week 48, n = 13, 8, 0 | 62.5 (27.5) | 78.1 (27.3) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Social Functioning, Week 72, n = 10, 7, 1 | 77.5 (20.2) | 78.6 (15.7) | 25.0 (NA) — Data is available only for one participant. Therefore, there is no standard deviation.
  Social Functioning, Week 96, n = 0, 6, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 83.3 (17.1) | NA (NA) — No participants were available for analysis in this arm at Week 96.
  Role Functioning -Emotional,Baseline,n =22, 18, 15 | 71.2 (38.9) | 62.0 (42.7) | 53.3 (45.1)
  Role Functioning-Emotional, Week 24, n=17, 13, 8 | 43.1 (43.7) | 20.5 (37.4) | 45.8 (50.2)
  Role Functioning - Emotional, Week 48, n= 13, 8, 0 | 43.6 (39.4) | 54.2 (46.9) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Role Functioning - Emotional, Week 72, n= 10, 7, 1 | 56.7 (49.8) | 81.0 (37.8) | 0.0 (0.0)
  Role Functioning - Emotional, Week 96, n = 0, 5, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 60.0 (43.5) | NA (NA) — No participants were available for analysis in this arm at Week 96.
  Mental Health, Baseline, n = 21, 18, 15 | 71.6 (18.1) | 62.9 (22.0) | 62.1 (20.8)
  Mental Health, Week 24, n = 17, 11, 8 | 58.8 (21.5) | 46.2 (18.6) | 62.0 (19.9)
  Mental Health, Week 48, n = 13, 8, 0 | 57.4 (24.0) | 61.0 (16.8) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Mental Health, Week 72, n = 9, 7, 1 | 66.7 (24.0) | 66.9 (17.8) | 36.0 (NA) — Data is available only for one participant. Therefore, there is no standard deviation.
  Mental Health, Week 96, n = 0, 6, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 58.3 (15.1) | NA (NA) — No participants were available for analysis in this arm at Week 96.
  Reported Health Transition,Baseline, n =22, 19, 15 | 3.0 (1.1) | 2.9 (0.9) | 3.3 (1.0)
  Reported Health Transition, Week 24, 17, 13, 9 | 3.8 (1.0) | 3.5 (1.2) | 3.2 (1.1)
  Reported Health Transition, Week 48, n = 13, 8, 0 | 2.9 (1.1) | 2.9 (1.1) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Reported Health Transition, Week 72, n = 10, 7, 1 | 2.8 (1.2) | 2.6 (1.3) | 4.0 (NA) — Data is available only for one participant. Therefore, there is no standard deviation.
  Reported Health Transition, Week 96, n = 0, 6, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 2.0 (0.9) | NA (NA) — No participants were available for analysis in this arm at Week 96.

13. Secondary Outcome: Mean Fatigue Severity Scale Scores for Groups A1, B1 and C Over Time (Part 2)
Description: The FSS is an instrument consisting of 10 self-administered questions. The FSS items were scored by calculating the average response to all answered items (including the 9 questions and the fatigue symptoms). Each of the 9 questions had answers within a score range of 1-7. A score of 1 for any question indicates less fatigue in everyday life and a score of 7 indicates a higher likelihood of fatigue in everyday life. The mean FSS scores are presented at Baseline (Day 1), Week 24, Week 48 and Week 72 (for Groups A1, B1 and C) and at Week 96 (for Groups B1 and C).
Time Frame: Baseline (Day 1), Week 24, Week 48 and Week 72, and Week 96
Population: The ITT population included all participants randomized and allocated to receive treatments. Here, 'n' = the number of participants analyzed for a given time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2)
Number analyzed (Participants) | 22 | 17 | 15
scores on a scale
  Baseline, n = 22, 17, 15 | 3.7 (1.6) | 3.8 (2.0) | 3.9 (1.9)
  Week 24, n = 17, 15, 9 | 4.2 (1.7) | 4.9 (1.6) | 4.8 (1.6)
  Week 48, n = 11, 7, 0 | 4.0 (1.5) | 4.5 (1.3) | NA (NA) — No participants were available for analysis in this arm at Week 48.
  Week 72, n = 8, 7, 1 | 3.9 (1.9) | 3.8 (2.2) | 5.3 (NA) — Data is available only for one participant. Therefore, there is no standard deviation.
  Week 96, n = 0, 7, 0 | NA (NA) — No participants were available for analysis in this arm at Week 96. | 4.5 (1.9) | NA (NA) — No participants were available for analysis in this arm at Week 96.

14. Secondary Outcome: Number of Participants With Fibrosis Grades 0 to 4 at Baseline (Part 2)
Description: Liver fibrosis stage was based upon biopsy and scored using the METAVIR system (Grade 0 to 4). Grade 0 indicates no fibrosis, Grade 1 indicates stellate enlargement of portal tract but without septa formation, Grade 2 indicates enlargement of portal tract with rare septa formation, Grade 3 indicates numerous septa without cirrhosis and grade 4 indicates cirrhosis. The number of participants with fibrosis grades ranging from 0 to 4 at Baseline (Day 1) is presented.
Time Frame: Baseline (Day 1)
Population: The ITT population included all participants randomized and allocated to receive treatments.
Measure: Number; unit: Number of participants
Groups:
- PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2): Eligible participants were administered PEG-IFN alfa-2a at a dose of 180 mcg SC once weekly for a total of 48 weeks and also received ribavirin at a dosage of 1,000 mg/day (for participants with a body weight </= 75 kg) or 1,200 mg/day (for participants with a body weight > 75 kg) orally for a total of 48 weeks. Participants with a positive HCV RNA level at Week 4 (>/= 15 IU/ml, TaqMan HCV Test) and negative HCV RNA level at Week 8 (</= 15 IU/ml, TaqMan HCV Test) were assigned to Group E. Participants had a treatment-free follow-up period of 24 weeks.
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2)
Number analyzed (Participants) | 25 | 17 | 15 | 23 | 26
Number of participants
  Grade 0 | 5 | 4 | 1 | 4 | 3
  Grade 1 | 6 | 3 | 2 | 8 | 9
  Grade 2 | 4 | 4 | 6 | 10 | 8
  Grade 3 | 5 | 2 | 5 | 1 | 1
  Grade 4 | 5 | 4 | 1 | 0 | 5

15. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events (Part 2)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 96
Population: as for outcome 7
Measure: Number; unit: Number of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2) | PEG-IFN Alfa-2a + Ribavirin (Not Assigned) (Part 2)
Number analyzed (Participants) | 36 | 25 | 20 | 42 | 45 | 8
Number of participants
  Number of participants with any AE | 36 | 25 | 19 | 40 | 43 | 7
  Number of participants with any SAE | 1 | 3 | 2 | 5 | 7 | 1

ADVERSE EVENTS:
Time Frame: Up to Week 96
Description: Adverse event data was reported for the safety population which included all participants who received at least on dose of (either) study drug (PEG-IFN alfa-2a or ribavirin) and had at least one post-baseline safety assessment.
Arm/Group | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1) | PEG-IFN Alfa-2a + Ribavirin (Not Randomized) (Part 1) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2) | PEG-IFN Alfa-2a + Ribavirin (Not Assigned) (Part 2)
Serious Adverse Events (participants affected / at risk) | 22/142 | 28/152 | 8/78 | 14/156 | 2/12 | 1/36 | 3/25 | 2/20 | 5/42 | 7/45 | 1/8
Other Adverse Events (participants affected / at risk) | 139/142 | 147/152 | 76/78 | 150/156 | 9/12 | 36/36 | 25/25 | 19/20 | 40/42 | 42/45 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) (N=142) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) (N=152) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) (N=78) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1) (N=156) | PEG-IFN Alfa-2a + Ribavirin (Not Randomized) (Part 1) (N=12) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) (N=36) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) (N=25) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) (N=20) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2) (N=42) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2) (N=45) | PEG-IFN Alfa-2a + Ribavirin (Not Assigned) (Part 2) (N=8)
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cryoglobulinaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basedow's Disease (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia Repair (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Cystectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pregnancy Of Partner (Social circumstances) | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mononeuritis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A) (Part 1) (N=142) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B) (Part 1) (N=152) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 1) (N=78) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 1) (N=156) | PEG-IFN Alfa-2a + Ribavirin (Not Randomized) (Part 1) (N=12) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group A1) (Part 2) (N=36) | PEG-IFN Alfa-2a + Ribavirin 72 Weeks (Group B1) (Part 2) (N=25) | PEG-IFN Alfa-2a + Ribavirin 24/72 Weeks (Group C) (Part 2) (N=20) | PEG-IFN Alfa-2a + Ribavirin 24 Weeks (Group D) (Part 2) (N=42) | PEG-IFN Alfa-2a + Ribavirin 48 Weeks (Group E) (Part 2) (N=45) | PEG-IFN Alfa-2a + Ribavirin (Not Assigned) (Part 2) (N=8)
Fatigue (General disorders) | 86 | 94 | 35 | 72 | 4 | 20 | 14 | 11 | 21 | 30 | 1
Influenza Like Illness (General disorders) | 60 | 57 | 41 | 61 | 5 | 15 | 14 | 7 | 13 | 14 | 1
Pyrexia (General disorders) | 29 | 34 | 9 | 14 | 2 | 5 | 5 | 0 | 6 | 7 | 0
Asthenia (General disorders) | 4 | 8 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Chills (General disorders) | 4 | 5 | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 1
Chest Pain (General disorders) | 4 | 2 | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 2 | 0
Irritability (General disorders) | 2 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Injection Site erythema (General disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Application Site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 35 | 39 | 15 | 24 | 2 | 6 | 7 | 1 | 5 | 7 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 27 | 19 | 18 | 2 | 6 | 5 | 3 | 8 | 13 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 29 | 39 | 8 | 27 | 0 | 4 | 3 | 1 | 7 | 7 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 17 | 31 | 8 | 19 | 1 | 7 | 6 | 2 | 1 | 8 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 11 | 12 | 0 | 6 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 5 | 16 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 4 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 30 | 44 | 20 | 27 | 0 | 7 | 1 | 1 | 5 | 7 | 1
Insomnia (Psychiatric disorders) | 16 | 24 | 9 | 16 | 1 | 5 | 3 | 0 | 5 | 5 | 0
Sleep Disorder (Psychiatric disorders) | 19 | 27 | 8 | 13 | 1 | 2 | 2 | 0 | 1 | 2 | 0
Depressed Mood (Psychiatric disorders) | 7 | 7 | 3 | 8 | 0 | 3 | 0 | 0 | 4 | 1 | 0
Aggression (Psychiatric disorders) | 5 | 8 | 4 | 3 | 1 | 1 | 0 | 1 | 0 | 3 | 0
Panic Attack (Psychiatric disorders) | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Affect Lability (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Libido Decreased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 27 | 22 | 11 | 15 | 0 | 10 | 3 | 2 | 7 | 7 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 20 | 16 | 11 | 23 | 1 | 1 | 1 | 0 | 4 | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 18 | 3 | 13 | 0 | 4 | 1 | 2 | 4 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 14 | 1 | 6 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 7 | 1 | 7 | 2 | 2 | 1 | 1 | 2 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 6 | 11 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 8 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 3 | 5 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 5 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 5 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 32 | 33 | 9 | 23 | 0 | 7 | 5 | 3 | 3 | 10 | 1
Leukopenia (Blood and lymphatic system disorders) | 31 | 20 | 11 | 19 | 0 | 3 | 2 | 0 | 1 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 15 | 4 | 3 | 0 | 2 | 2 | 0 | 4 | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 8 | 2 | 3 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 5 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 24 | 12 | 21 | 0 | 8 | 6 | 2 | 4 | 8 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 25 | 10 | 13 | 3 | 4 | 2 | 0 | 3 | 3 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 3 | 4 | 0 | 2 | 2 | 3 | 1 | 3 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 0 | 9 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 1 | 4 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 27 | 10 | 13 | 0 | 7 | 6 | 2 | 3 | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 23 | 8 | 16 | 0 | 6 | 3 | 0 | 2 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 9 | 2 | 6 | 0 | 0 | 1 | 1 | 4 | 3 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 9 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 16 | 26 | 6 | 22 | 0 | 10 | 3 | 3 | 4 | 4 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 17 | 16 | 9 | 17 | 0 | 3 | 1 | 1 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 19 | 17 | 8 | 7 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Appetite Disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 42 | 38 | 10 | 26 | 1 | 8 | 3 | 5 | 8 | 10 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 16 | 23 | 6 | 9 | 0 | 2 | 1 | 1 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 5 | 14 | 5 | 7 | 0 | 2 | 1 | 0 | 4 | 2 | 0
Influenza (Infections and infestations) | 5 | 7 | 2 | 5 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 3 | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 3 | 0
Oral Herpes (Infections and infestations) | 4 | 5 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 7 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 2 | 6 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulpitis Dental (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 8 | 23 | 4 | 8 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 7 | 10 | 3 | 6 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 16 | 20 | 8 | 9 | 0 | 3 | 2 | 1 | 1 | 1 | 0
Weight Decreased (Investigations) | 17 | 14 | 3 | 9 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Visual Impairment (Eye disorders) | 4 | 8 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 3 | 6 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Dry Eye (Eye disorders) | 3 | 3 | 1 | 3 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Abnormal Sensation In Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiovascular Disorder (Cardiac disorders) | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.